CLINICAL TRIAL: NCT07007754
Title: Effects of Voice Records on Vital Signs, Pain and Serum Cortisol Levels in Surgical Intensive Care Unit: Randomized-controlled Study
Brief Title: Effects of Voice Records on Patient Outcomes Surgical Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ezgi Arslan, PhD, Research Assisstant (Principal Investigator), Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Voice Record
Record Dates: First submitted 2025-05-12; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Intensive Care Unit Patients; Pain Management; Stress Response
Keywords: Abdominal surgery; intensive care unite; nursing care; voice record
MeSH Terms: conditions — Agnosia; Fractures, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Family voice records (Experimental): In addition to the general care provided by health professionals in ICU, the intervention group-1 listen to family voice records.
  Interventions: Procedure: Voice recording playback
- Notr voice record (Experimental): In addition to the general care provided by health professionals in ICU, the intervention group-1 listen to nötr voice records.
  Interventions: Procedure: Voice recording playback
- Control group (No Intervention): The control group received general care provided by healthcare professionals in the ICU.

INTERVENTIONS:
Procedure: Voice recording playback — Voice recordings were created from a text containing 12 standardised messages common to both the patient's relatives and the researcher and expert opinion was obtained in terms of the applicability of the created text. Before the intervention, the postoperative patient's suitability was determined by the patient's statement and the researcher's observations. No intervention was performed if the patient had nausea/vomiting, pain or agitation before the intervention. Kingboss 8 Gb+ 650 hours uninterrupted digital voice recorder and headphones were used for voice recording. When the voice recorder and headphones were to be used in a different patient, they were wiped with 70% alcohol and used after waiting for 2 minutes in accordance with the manufacturer's instructions. The voice of one of the family members was recorded for Intervention group-1 patients and the voice of one of the researchers was (nötr voice) recorded for intervention group-2.
  Arms: Family voice records; Notr voice record

SUMMARY:
This randomized kontrolled study is aimed to contribute to the literature on recognising, evaluating and reducing stress in the intensive care unit, which is one of the main responsibilities of surgical nurses, and to increase awareness on the subject.

DETAILED DESCRIPTION:
The condition of having surgery, the severity of the disease, being admitted to the intensive care unit in the postoperative period and the presence of many invasive interventions in the body, intense feelings of pain and fear, loss of autonomy, helplessness, and fear of death create a heavy physical, psychological and emotional burden on patients undergoing surgery. All these factors increase the stress level in the patient by causing many metabolic and hormonal changes, and as a result of this stress response, negative conditions such as hyperglycaemia, delay in recovery, and decreased immunity can be seen.

Nurses have main roles and responsibilities in intensive care settings such as caring for patients, participating in treatment, informing and counselling patients and their relatives. Within the scope of these roles and responsibilities, nurses should be aware of the stress experienced by patients, recognise the factors that may cause stress, plan, implement and evaluate basic nursing interventions such as increasing coping strategies and social support in the management and alleviation of stress, informing and counselling, increasing the patients orientation, and enabling the patient to participate in care in order to reduce the level of stress experienced by patients and protect their physical and biopsychosocial integrity.

There are no studies in the literature examining the effects of listening to audio recordings, which is an easy, inexpensive and non-pharmacological intervention for stress management of patients in intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* To determined as being over 18 years of age,
* To staying in the ICU for at least two hours,
* To being hospitalised in the ICU for the first time,
* To being able to speak and understand Turkish.

Exclusion Criteria:

* To determined as being pregnant,
* To having a diagnosis of neurological/psychiatric disorder,
* To having hearing problems,
* To using cortisol-derived drugs,
* To having a disease that may affect serum cortisol level, exhibiting agitated behaviour and
* To experiencing intense nausea and vomiting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Pain level | Postoperative 1st, 2nd and 3rd days at 06:00 A. M.
  A numerical rating scale was used to evaluate the pain. The scale was marked from 0 to 10 based on the patient's self-report. 0 indicates no pain, while 10 points indicates unbearable pain.
Blood pressure | Postoperative 1st, 2nd and 3rd days at 06:00 A. M.
  Since the patients were monitored in the intensive care unit and invasive blood pressure measurements were performed, the values monitored on the Mindray patient monitor were added to the data collection form.
Serum cortisol level | Postoperative 1st, 2nd and 3rd days at 06:00 A. M.
  The serum cortisol level in the blood was reported in an independent private laboratory by taking a blood sample.
Blood glucose level | Postoperative 1st, 2nd and 3rd days at 06:00 A. M.
  The blood glucose level was assessed using Gluko Navi brand glucometer with fingertip measurement.
Hearth rate | Postoperative 1st, 2nd and 3rd days at 06:00 A. M.
  Since the patients were monitored in the intensive care unit and pulse rate was measured, the values monitored on the Mindray patient monitor were added to the data collection form.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Zafer Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 6 months after publication